CLINICAL TRIAL: NCT00436059
Title: The Efficacy of Velcade on Bone Tissue During Myelomatosis (Bone Marrow Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/175
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
The primary objective of the the study is to investigate the changes in bone remodeling during Velcade treatment.

DETAILED DESCRIPTION:
20 patients will be included in the study over a 2 year period. Before, during and after treatment we will measure NTX-I, CTX-I, CTX-MMP, bALP, DKK-1, PINP, TRAcP and PTH. NTX, CTX and CTX-MMP are measured to estimate bone degradation. TRAcP is measured to estimate the activity of the osteoclasts. bALP and DKK-1 is measured to evaluate the activity of the osteoblasts and PINP is measured as a marker of new bone formation. PTH is measured in order to evaluate if the positive effects that is observed in bone formation in relations to velcade treatment is due to the pulsative way velcade is administered.

The effect of the velcade treatment will be evaluated by x-ray, bone marrow and m-component.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated multiple myeloma

Exclusion Criteria:

* Use of bisfosfonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes in bone markers during treatment

SECONDARY OUTCOMES:
Changes in osteolysis during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Torben Plesner, MD, Principal Investigator — Vejle Hospital
Locations (2):
- Denmark (2):
  - University Hospital Odense, Odense, Odense
  - Vejle Hospital, Vejle, Vejle